CLINICAL TRIAL: NCT00359957
Title: Activity, Diet, and Visceral Adiposity: New Care Emerging (ADVANCE) Project
Brief Title: Efficacy of Increasing Physical Activity to Reduce Children's Visceral Fat
Acronym: ADVANCE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Brian Saelens, PhD, Children's Hospital and Regional Medical Center, Seattle
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK60476 (completed); NIH/NIDDK K23 DK60476
Record Dates: First submitted 2006-08-01; First posted 2006-08-03 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Obesity
Keywords: Pediatric obesity; Physical activity; Visceral fat; Weight
MeSH Terms: conditions — Obesity; Pediatric Obesity; Motor Activity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ADDED condition - behavioral intervention for modifying diet and physical activity, with greater emphasis on physical activity than the STANDARD condition
  Interventions: Behavioral: Pediatric Obesity Intervention + High Activity (ADDED)
- 2 (Active Comparator): STANDARD condition - behavioral intervention for modifying diet, with little emphasis on physical activity
  Interventions: Behavioral: Pediatric Obesity Intervention (STANDARD)

INTERVENTIONS:
Behavioral: Pediatric Obesity Intervention (STANDARD) — 14 weekly behavioral intervention visits with parent and child; individual family sessions (25-30 minutes) and separate parent and child groups (40 minutes)
  Arms: 2
Behavioral: Pediatric Obesity Intervention + High Activity (ADDED) — 14 weekly behavioral intervention visits with parent and child; individual family sessions (25-30 minutes) and separate parent and child groups (40 minutes)
  Arms: 1

SUMMARY:
The purpose of this trial is to examine whether adding greater physical activity to standard family-based behavioral pediatric obesity treatment decreases the amount of visceral fat among treated overweight children.

DETAILED DESCRIPTION:
Adult studies suggest that greater visceral fat confers more health risk than peripheral fat accumulation and that physical activity interventions (as part of general weight control interventions) are efficacious in reducing adults' visceral fat. There are few studies examining the impact of physical activity and/or general weight loss on children's visceral fat accumulation. The present study compares standard family-based behavioral weight control treatment for pediatric obesity (STANDARD) with standard treatment plus added emphasis on participants attaining high levels of physical activity (ADDED). Both conditions receive the same behavioral dietary intervention and therapeutic contact and attention. The ADDED condition receives the recommendation and goal to be active at least 90 minutes per day, with behavioral strategies targeting increasing and sustaining these high levels of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* 7-12 years old
* >85th percentile BMI
* have at least one parent with a BMI>25
* able to engage in at least moderate intensity physical activity
* child and parent willing and able to participate in behavioral treatment
* English-speaking

Exclusion Criteria:

* child or parent already enrolled in another weight control program
* child or parent with a medical condition known to affect weight or growth
* child or parent with significant mental illness that would interfere with engaging in treatment
* child or parent with a current or past diagnosed eating disorder
* child or parent currently taking any medication that affects weight or growth
* child who is more than 120% above their median BMI for age and gender

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Visceral adiposity | Change over 3-4 month period

SECONDARY OUTCOMES:
Subcutaneous abdominal adiposity | Change over 3-4 month period
Total body fat | Change over 3-4 month period
Body mass index | Change over 3-4 month period
Physical activity | Change over 3-4 month period

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Saelens, Ph.D., Principal Investigator — Children's Hospital and Regiona Medical Center, Seattle
Locations (1):
- Children's Hospital and Regional Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Saelens BE, Grow HM, Stark LJ, Seeley RJ, Roehrig H. Efficacy of increasing physical activity to reduce children's visceral fat: a pilot randomized controlled trial. Int J Pediatr Obes. 2011 Apr;6(2):102-12. doi: 10.3109/17477166.2010.482157. Epub 2010 Jun 7. PMID 20528109